CLINICAL TRIAL: NCT07265232
Title: Real World Clinical Effectiveness & Safety of Vesemnogene Lantuparvovec for Spinal Muscular Atrophy (SMA) in Low-middle Income Countries (LMIC).
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lantu Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR 25-02
Record Dates: First submitted 2025-11-21; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Spinal Muscular Atrophy (SMA)
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The selected dose inchildren ≥ 6 months of age (Experimental): Administration the selected dose of Vesemnogene Lantuparvovec in children > 6 months of age
  Interventions: Biological: vesemnogene lantuparvovec

INTERVENTIONS:
Biological: vesemnogene lantuparvovec — Exploratory study evaluating the safety and efficacy of vesemnogene lantuparvovec in patients with SMA.

SUMMARY:
The study objective is to determine the real-world safety and effectiveness of Vesemnogene lantuparvovec for the treatment of SMA.

The specific objectives are:

* To determine clinical effectiveness of Vesemnogene lantuparvovec therapy for SMA as evaluated by developmental gross motor milestone and survival.
* To describe the safety profile of Vesemnogene therapy for SMA as evaluated by adverse events reporting and laboratory tests, and monitoring of Adverse events of special interest.

DETAILED DESCRIPTION:
This is an observational study designed to determine the real-world safety and effectiveness of Vesemnogene lantuparvovec therapy for SMA. Potential patients with genetic diagnosis of SMA will be evaluated for eligibility to undergo available gene therapies. Following the administration of Vesemnogene therapy, patient will be monitored for toxicity and response to treatment. No subjects will be withdrawn from the study, and subjects could freely drop out from the study anytime, simply by not showing up.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Genetic confirmation of SMA (biallelic deletion or mutation of SMN1).
3. SMA clinical phenotype and condition, that in the opinion of the treating physician, treatment with Vesemnogene will likely be beneficial.
4. Absence of contraindications for spinal tap procedure or administration of intrathecal therapy.
5. Total AAV antibody titres < 1:20 as determined by ELISA assay.
6. Normal liver function (AST/ALT < 3XULN, Bilirubin <3.0 mg/dL).
7. Unable to access or failure to respond to currently available curative treatments for SMA.

Exclusion Criteria:

None

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2030-10-15 (Estimated); Study Completion 2030-10-15 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with adverse events (AEs), serious adverse events (SAEs) | Baseline up to 5 years old
  Participants are monitored for safety from baseline up to the end of the follow-up period.

SECONDARY OUTCOMES:
Change from baseline in developmental gross motor milestones achieved according to WHO criteria | Baseline up to 5 years old
  For patients with SMA, the percentage of participants who are able to preserve ambulatory function.
Event-free Survival until the 5th year or the last follow-up | Baseline up to 5 vears old
  Event-free survival was defined as the number of participants who did not die, did not require permanent ventilation and did not withdraw from the study until the 5th year or the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Tzu chi hospital, Jakarta, Indonesia, Indonesia